CLINICAL TRIAL: NCT02151812
Title: A Prospective Randomized Multicenter Non-inferiority Clinical Study to Determine the Safety and Performance of the Agent™ Paclitaxel-Coated PTCA Balloon Catheter (Hemoteq) Compared to the SeQuent® Please Paclitaxel-Releasing Coronary Balloon Catheter (B.Braun) for the Treatment of Coronary In-Stent Restenosis (AGENT-ISR)
Brief Title: Comparison of Agent™ and SeQuent® Please Paclitaxel Coated Balloon Catheters in Coronary In-stent Restenosis (AGENT-ISR)
Acronym: AGENT-ISR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hemoteq AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HTQ002-Agent-ISR; CIV-13-11-011728 (Other: EUDAMED)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Coronary Artery Disease; Coronary Restenosis; Coronary Atherosclerosis; Coronary Arteriosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Agent Paclitaxel-coated balloon (Experimental): drug-coated balloon dilatation of the index lesion using a single Agent(TM) balloon that completely covers the restenotic lesion
  Interventions: Device: Agent Paclitaxel-coated balloon
- SeQuent Please Paclitaxel-coated balloon (Active Comparator): drug-coated balloon dilatation of the index lesion using a single SeQuent(R) Please balloon that completely covers the restenotic lesion
  Interventions: Device: SeQuent® Please Paclitaxel-coated Balloon

INTERVENTIONS:
Device: Agent Paclitaxel-coated balloon — After successful pre-dilatation, the index lesion is dilated with a single drug-coated balloon that completely covers the restenotic lesion.
  Arms: Agent Paclitaxel-coated balloon
Device: SeQuent® Please Paclitaxel-coated Balloon — After successful pre-dilatation, the index lesion is dilated with a single drug-coated balloon that completely covers the restenotic lesion.
  Arms: SeQuent Please Paclitaxel-coated balloon

SUMMARY:
The primary objective of this study is determine the safety and performance of the Agent™ Paclitaxel-Coated PTCA Balloon Catheter compared to the SeQuent® Please Paclitaxel-Releasing Coronary Balloon Catheter for the treatment of patients with narrowed previously-stented coronary arteries (in-stent restenosis).

The performance will be determined at six months post-procedure by quantitative coronary angiography (QCA) to measure Late Lumen Loss (LLL) in the re-opened stented segment. QCA results will be assessed by an independent, blinded angiographic core lab.

Study statistical hypothesis: The loss of in-stent luminal diameter at six months after treatment of the restenosed stent with the Agent™ study device is not larger than the respective LLL after treatment with the SeQuent® Please control devices, i.e. study device is non-inferior to the control device with respect to LLL.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age
* Subject is willing and able to provide informed consent
* Subject is eligible for percutaneous coronary intervention
* Subject is willing to comply with all protocol-required follow-up evaluations
* Women of child-bearing potential must agree to use a reliable method of contraception
* In-stent restenosis in a lesion previously treated with either a drug-eluting or bare metal stent, located in a native coronary artery with a reference vessel diameter ≥ 2.0 mm and ≤ 3.5 mm
* Target lesion length must be ≤ 28 mm (by visual estimate) and must be covered by only one balloon
* Target lesion must have visually estimated stenosis ≥ 70% and < 100% in asymptomatic patients
* Target lesion must have visually estimated stenosis ≥ 50% and < 100% in symptomatic patients
* Thrombolysis in Myocardial Infarction (TIMI) grade flow in the target lesion must be ≥ 1
* Target lesion must be successfully pre-dilated.

Exclusion Criteria:

* Patient has life expectancy of less than 24 months
* Patient with known coronary artery spasm
* Patient with unprotected left main coronary artery disease
* Patient has current problems with substance abuse
* Patient has planned procedure that may cause non-compliance with the protocol or confound data interpretation
* Patient is participating in another investigational drug or device clinical study that has not reached its primary endpoint
* Patient intends to participate in another investigational drug or device clinical study within 12 months after the index procedure
* Woman who is pregnant or nursing
* Left ventricular ejection fraction < 25%
* Patient had PCI or other coronary interventions within the last 30 days
* Planned PCI or CABG after the index procedure
* Patient to receive other PCI interventions in the target vessel, such as rotablation, laser atherectomy, cutting balloon, DCB, DES, BMS, bioabsorbable scaffold etc.
* Patient to receive DCB in non-target coronary vessels
* Acute MI < 72h
* Cardiogenic shock
* Known allergies against Paclitaxel or other components of the used medical devices
* Known hypersensitivity or contraindication for contrast dye that cannot be adequately pre-medicated
* Intolerance to antiplatelet drugs, anticoagulants required for the procedure
* Platelet count < 100k/mm3 or > 500k/mm3
* Patient with renal failure with a serum creatinine of > 2.5mg/dL who is receiving dialysis or chronic immunosuppressant therapy
* Target lesion is located within a bifurcation involving a major side branch > 2 mm in diameter
* Target lesion is located within a saphenous vein graft or an arterial graft
* Target lesion with TIMI grade flow = 0 (total occlusion)
* Thrombus present in the target vessel
* > 50% stenosis of an additional lesion proximal or distal to the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2014-08-13 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
in-stent late lumen loss | six months
  In-stent late lumen loss (LLL) of the treated stented segment after PTCA using the Agent(TM) study device in comparison to the LLL after PTCA using the SeQuent(R) Please control device as measured by QCA at six months post-index procedure.

SECONDARY OUTCOMES:
technical success rate | during index procedure, less 1 hour
  The ability to cross and dilate the lesion to achieve residual angiographic stenosis no greater than 30 percent
clinical procedural success rate | within 24 hours of index procedure
  Technical success with no composite of all death and MI noted within 24 hours of the index procedure.
In-stent percent diameter stenosis | 6 months post-index procedure
  In-stent percent diameter reduction measured within the borders of the stent
In-segment percent diameter stenosis | 6 months post-index procedure
  In-segment percent diameter reduction measured in the stented segment plus 5mm on either side.
In-stent binary restenosis rate | 6 months post-index procedure
  In-stent binary restenosis is defined as ≥50% luminal narrowing within the borders of the stent observed at follow-up QCA.
In-segment binary restenosis rate | 6 months post-index procedure
  In-segment binary restenosis is defined as ≥50% luminal narrowing in the stented segment plus 5mm on either side observed at follow-up QCA.
In-segment late lumen loss | 6 months post-index procedure
  In-segment late lumen loss is the in-segment minimal lumen diameter (MLD) post index procedure minus the in-segment MLD at 6 months follow-up as determined by QCA.
In-stent minimal lumen diameter (MLD) | 6 months post-index procedure
  In-stent MLD is measured within the borders of the stent.
In-segment minimal lumen diameter (MLD) | 6 months post-index procedure
  In-segment MLD is measured in the stented segment plus 5mm on either side.
Target lesion revascularization (TLR) rate | pre-discharge, estim. <10 days
  TLR rate during index in-hospital stay
Target lesion revascularization (TLR) rate | 30 days
Target lesion revascularization (TLR) rate | six months
Target lesion revascularization (TLR) rate | 12 months
Target lesion revascularization (TLR) rate | 24 months
Target lesion revascularization (TLR) rate | 36 months
Target vessel revascularization (TVR) rate | pre-discharge, estim. <10 days
  TVR rate during index in-hospital stay
Target vessel revascularization (TVR) rate | 30 days
Target vessel revascularization (TVR) rate | six months
Target vessel revascularization (TVR) rate | 12 months
Target vessel revascularization (TVR) rate | 24 months
Target vessel revascularization (TVR) rate | 36 months
Cardiac, non-cardiac and all death rates | pre-discharge, estim. <10 days
  rates during index in-hospital stay
Cardiac, non-cardiac and all death rates | 30 days
Cardiac, non-cardiac and all death rates | six months
Cardiac, non-cardiac and all death rates | 12 months
Cardiac, non-cardiac and all death rates | 24 months
Cardiac, non-cardiac and all death rates | 36 months
Myocardial infarction rates (by 3rd Universal Definition: all MI, QWMI, NQWMI) | pre-discharge, estim. <10 days
  rates during index in-hospital stay
Myocardial infarction rates (by 3rd Universal Definition: all MI, QWMI, NQWMI) | 30 days
Myocardial infarction rates (by 3rd Universal Definition: all MI, QWMI, NQWMI) | six months
Myocardial infarction rates (by 3rd Universal Definition: all MI, QWMI, NQWMI) | 12 months
Myocardial infarction rates (by 3rd Universal Definition: all MI, QWMI, NQWMI) | 24 months
Myocardial infarction rates (by 3rd Universal Definition: all MI, QWMI, NQWMI) | 36 months
Stent thrombosis rate (by ARC definition) | pre-discharge, estim. <10 days
  rates during index in-hospital stay
Stent thrombosis rate (by ARC definition) | 30 days
Stent thrombosis rate (by ARC definition) | six months
Stent thrombosis rate (by ARC definition) | 12 months
Stent thrombosis rate (by ARC definition) | 24 months
Stent thrombosis rate (by ARC definition) | 36 months
Target lesion failure (TLF) rate (composite of cardiac death, MI and TLR) | pre-discharge, estim. <10 days
  rates during index in-hospital stay
Target lesion failure (TLF) rate (composite of cardiac death, MI and TLR) | 30 days
Target lesion failure (TLF) rate (composite of cardiac death, MI and TLR) | six months
Target lesion failure (TLF) rate (composite of cardiac death, MI and TLR) | 12 months
Target lesion failure (TLF) rate (composite of cardiac death, MI and TLR) | 24 months
Target lesion failure (TLF) rate (composite of cardiac death, MI and TLR) | 36 months
Target vessel failure (TVF) rate (composite of cardiac death, MI and TVR) | pre-discharge, estim. <10 days
  rates during index in-hospital stay
Target vessel failure (TVF) rate (composite of cardiac death, MI and TVR) | 30 days
Target vessel failure (TVF) rate (composite of cardiac death, MI and TVR) | six months
Target vessel failure (TVF) rate (composite of cardiac death, MI and TVR) | 12 months
Target vessel failure (TVF) rate (composite of cardiac death, MI and TVR) | 24 months
Target vessel failure (TVF) rate (composite of cardiac death, MI and TVR) | 36 months
Change in Quality of Life | six months
  Functional status of general health-related quality of life (QoL) measured by changes in SF-12 scores and EQ5D scores as compared to baseline
Change in Quality of Life | 12 months
  Functional status of general health-related quality of life (QoL) measured by changes in SF-12 scores and EQ5D scores as compared to baseline
Change in Quality of Life | 24 months
  Functional status of general health-related quality of life (QoL) measured by changes in SF-12 scores and EQ5D scores as compared to baseline
Change in Quality of Life | 36 months
  Functional status of general health-related quality of life (QoL) measured by changes in SF-12 scores and EQ5D scores as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christian W. Hamm, MD, Principal Investigator — University Giessen, Germany
Locations (12):
- France (5):
  - Centre Hospitalier Saint Joseph Saint Luc de Lyon, Lyon
  - Clinique du Millénaire, Montpellier, Montpellier
  - CHU Montpellier, Hôpital Arnaud de Villeneuve, Montpellier
  - CHU de Nantes, Hopital Laennec, Nantes
  - Clinique Saint Hilaire, Rouen, Rouen
- Germany (7):
  - Kerckhoff-Klinik, Bad Nauheim
  - Charité Universitaetsmedizin Berlin, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - University Giessen, Giessen
  - Klinikum Am Steinenberg, Reutlingen
  - Universitaetsklinikum Rostock, Rostock
  - Universitaetsklinikum Ulm, Ulm

REFERENCES:
- [Derived] Hamm CW, Dorr O, Woehrle J, Krackhardt F, Ince H, Zeus T, Berland J, Piot C, Roubille F, Schult I, Allocco DJ, Nef H. A multicentre, randomised controlled clinical study of drug-coated balloons for the treatment of coronary in-stent restenosis. EuroIntervention. 2020 Jul 17;16(4):e328-e334. doi: 10.4244/EIJ-D-19-00051. PMID 31746743